CLINICAL TRIAL: NCT02927743
Title: Effect of Continuous Evidence-based Feed Back to Increase Appropriate Use of Antibiotics
Brief Title: Effect of Evidence-based Reminders on Use of Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloria Cristina Cordoba (Other)
Collaborators: Society of Family Medicin La Paz-Bolivia (Unknown); University of Itapua, Paraguay (Unknown); University of the Republic, Uruguay (Other); Society of General and Family practice, Misiones- Argentina (Unknown)
Responsible Party: Sponsor-Investigator, Gloria Cristina Cordoba, MD-MPH, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HAPPY-AUDIT II/cRCT
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Infections; Antibiotics
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- evidence-based online feedback (Active Comparator): During three months GPs will receive weekly feedback about evidence-based management of respiratory tract infections. In order to control that they read the material, there is a questionnaire, they have to fill in every week
  Interventions: Behavioral: evidence-based online feedback
- control (No Intervention): GPs will register data without receiving online feed-back

INTERVENTIONS:
Behavioral: evidence-based online feedback — GPs received during three months weekly mails about evidence-based practice and a small questionnaire to reflect about their practice and the new knowledge
  Arms: evidence-based online feedback

SUMMARY:
Inappropriate use of antibiotics in primary care is associated with Development of antibiotic resistant strains. As part of a quality improvement program carried out in primary care in Uruguay, Argentina, Paraguay and Bolivia, a cluster randomized control trial was performed. The aim of the study was to assess whether the use of continuous evidence-based feedback about management of respiratory tract infections could decrease use of antibiotics in Acute bronchitis, common cold and acute otitis media.

DETAILED DESCRIPTION:
Excessive and inappropriate use of antibiotics is one of the most important reasons for development of resistant bacteria.

One of the key strategies to curb the development of antibiotic resistance is to promote intervention at primary care level as more than 90% of antibiotics are prescribed by general practitioners - especially in patients suffering from respiratory tract infections.

The main bacteria causing respiratory tract infections are S. pneumoniae y Haemophilus influenzae. The first one is associated with a significant increase in morbidity and mortality in Latin America.

Approximately 80% of respiratory tract infections have a viral cause, are harmless and self-limiting and in most cases patients recover without specific treatment. Antibiotic treatment is superfluous and in some cases even harmful because of side effects.

Infections caused by resistant bacteria leads to increased mortality, prolonged hospital stay and social collateral damage. Therefore, in 2013 the World Economic Forum pointed out antibiotic resistance as one of the three most important threats to economic and social development.

The World Health Organisation (WHO) launched in 20121 a global strategy to hold back antimicrobial resistance. According to this strategy "the battle against infectious diseases is far from being over. Not only do they continue to cause a large number of infections and deaths, particularly in developing countries, but the emergence and spread of antimicrobial resistance is now also threatening to undermine our ability to treat infections and save lives". The WHO has proposed a number of initiatives against the emergence of resistant bacteria, including interventions to promote proper use of antibiotics.

HAPPY AUDIT II (HA-II) - PART OF THE SOLUTION

HAPPY AUDIT - II is the second phase of HAPPY AUDIT - I, which was a project funded by the European Union to promote appropriate use of antibiotics in 6 countries with a very heterogeneous pattern of consumption of antibiotics and prevalence of resistant strains.

440 general practitioners registered data in winter 2008 and 2009. Inappropriate antibiotic use was reduced by 10% and in pathologies such as acute bronchitis, there was a 50% reduction in use of antibiotics.

In Argentina, 48 general practitioners participated in the whole process and reached a 30% reduction of unnecessary prescriptions of antibiotics in patients with acute bronchitis, sinusitis and pharyngitis.

The positive experience of the first phase has shown the importance and the potential to spread the project to other provinces of Argentina and other South American countries. Our prior knowledge will be used in the HAPPY AUDIT II SOUTH AMERICA to plan interventions for patients and GPs through the methodology APO (Audit Project Odense) which is based on:

1. self-reflection of physicians and group discussion on their prescription patterns,
2. patient education,
3. Development of a multi-faceted intervention.

The overall purpose of the project is to promote the rational use of antibiotics. This will be achieved through the following specific objectives:

1. Preparation of intervention materials for patients and professionals.
2. Implementation of APO cycles in 4 countries.
3. Initial registration of GPs and use of antibiotics for their RTI patients.
4. Analysis of the results of the first registration to identify quality problems in prescription.
5. Development of a multifaceted intervention.
6. Implementation of a cluster randomized control trial to assess the effect of the intervention.
7. Final registration to evaluate the effect of the intervention.

PROJECT ORGANIZATION

180 GPs will participate: Argentina 80 physicians, Bolivia 30 physicians, Paraguay 40 physicians and Uruguay 30 physicians.

The investigators will use the APO methodology, which based on a "bottom-up" approach seeks to change practice behaviour among GPs. The GPs voluntarily participate and set their own quality criteria in order to improve the quality of their own service.

The APO method includes:

* Initial registration of GPs own activities (3 weeks)
* Intervention (online evidence-based reminders during final registration)
* Final registration and evaluation (3 weeks)

Schedule 2014

February - May 2014 - coordinators and researchers first meeting

June - August 2014 - First audit registration during 15 days.

October 2014 - Coordinators and researchers second meeting

March 2015 - Meeting with General Practitioners from all provinces and/ or countries. This meeting will be divided into two parts:

1. Discussion of the results from the first registration;
2. Discussion about the use of quality indicators to decrease inappropriate use of antibiotics.

June - August 2015 - Second registration, intervention (online weekly feedback on evidence-based management of respiratory tract infections)

November 2016 - Assessment of the intervention.

April 2017 - Publication of results

ELIGIBILITY:
Inclusion Criteria:

* General practitioners working in primary care
* Patients with suspected respiratory tract infection

Exclusion Criteria:

* Patients that have already started an antibiotic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8053 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
20% difference in use of antibiotics in patients with suspected Acute bronchitis | 3 months

SECONDARY OUTCOMES:
20% difference in the use of antibiotics in suspected acute otitis media | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark